CLINICAL TRIAL: NCT00476944
Title: Minimizing Post-Procedural Vascular Complications: Comparing Bivalirudin Versus Heparin/GP IIB/IIA in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Comparing Bivalirudin Versus Heparin/ GP IIB/IIA in Patients Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gold, Herman K., MD (Individual)
Collaborators: The Medicines Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2006P000944
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease
Keywords: CAD; Coronary Artery Disease; Angiomax; Bivalirudin; PCI; MAVE; Heparin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI)

SUMMARY:
The purpose of this study is to compare the rates of vascular related complications in patients undergoing percutaneous coronary intervention assigned to one of two arms: 1) bivalirudin + provisional Gp IIB/IIIA use versus 2) heparin + Gp IIB/IIIA (eptifibatide (Integrilin®)) use.

DETAILED DESCRIPTION:
Anti-thrombotic therapies have enhanced the safety of percutaneous coronary intervention (PCI). In addition to aspirin, heparin and platelet glycoprotein (Gp) IIB/IIIA receptor inhibition have been used as the reference strategy to reduce the incidence of ischemic complications during coronary interventions 1. However, the success of this strategy is limited by increased bleeding risk, prolonged drug infusions (12 hours), and patient inconveniences (such as lying flat for hours until blood coagulation becomes normal and sheaths can be safely removed). Peri-procedural bleeding due to vascular complications is one of the most frequent complications of PCI and is associated with adverse events 2.

Newer anti-thrombotic strategies may further improve outcomes after PCI. The efficacy of a direct thrombin inhibitor bivalirudin (Angiomax™) was investigated in a randomized controlled clinical trial as a replacement for the strategy of heparin/Gp IIB/IIIA inhibition in patients undergoing coronary intervention. The REPLACE-2 study, which randomized over 6000 patients found short and long-term clinical outcomes with bivalirudin were as effective as heparin/Gp IIB/IIIA inhibition combination with evidence of significantly less major and minor bleeding 3, 4. This led to approval of the 0.75 mg/kg/1.75 mg/kg/hr dose of Angiomax® by the Food and Drug Administration for use as an anticoagulant in patients with unstable angina undergoing PCI.

It is now routinely accepted that early sheath removal after PCI reduces femoral access site complications and leads to earlier ambulation, earlier discharge, improved patient satisfaction 5. Heparin-based anticoagulation requires monitoring of the coagulation status to determine readiness for sheath removal because of the lack of predictable duration of anticoagulation with heparin. Because clearance of bivalirudin occurs mostly by proteolytic cleavage by thrombin, the drug has more predictable pharmacokinetics and exhibits linear dose relationship with respect to plasma concentrations and coagulation assay endpoints 6. Preliminary studies indicate sheath removal 2 hours after cessation of bivalirudin without coagulation monitoring is safe 5. While REPLACE-2 suggested that catheterization related vascular complications were decreased with bivalirudin, specific data on these endpoints and others such as time to ambulation and time to discharge were not collected because of the blinded nature of the trial. Currently the rate of vascular complications at MGH for patients undergoing PCI is 4.0% which significantly exceeds the national rate of 1.9% (95% CI 1.1 to 3.2) 7.

We will conduct a randomized clinical trial in patients undergoing PCI to compare the rates of vascular related complications between patients assigned to one of two arms: 1) bivalirudin + provisional Gp IIB/IIIA use versus 2) heparin + Gp IIB/IIIA (eptifibatide (Integrilin®)) use. The primary endpoint will be a composite of vascular related groin complications (MAVE-major adverse vascular endpoints as defined in next section). Secondary endpoints will be 1) time to sheath pull; 2) time to ambulation; and 3) occurrence of major and minor bleeding peri-catheterization.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

* The patients must be >18 years of age
* Patients must have been referred for percutaneous coronary intervention (PCI)
* Diagnosis of angina pectoris defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
* Treatment of lesions in native coronary vessels or bypass grafts requiring angioplasty or stenting.
* Patient is willing to comply with the specified follow-up evaluation;
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

* Patient has experienced an ST-segment elevation myocardial infarction within the preceding 24 hours.
* Active internal bleeding or bleeding diathesis, surgery, trauma, or gastrointestinal or genitourinary tract bleeding within past 6 weeks; prior intracranial bleeding; or platelet count<100,000
* Woman of child-bearing potential unless demonstrated negative pregnancy test
* End Stage Renal Disease requiring hemodialysis
* Recipient of heart transplant;
* Current treatment with 1) intravenous unfractionated heparin or treatment with low molecular weight heparin within past 8 hours; 2)bivalirudin; 3)abciximab; 4)eptifibatide; or tirofiban
* Ongoing need for warfarin or heparin therapy
* Known allergies to aspirin, clopidogrel bisulfate (Plavix®) and/or heparin;
* Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in an investigational drug or another device study;
* Any contraindication to glycoprotein IIb/IIIa inhibitor (eptifibatide (Integrilin®)) or bivalirudin therapy;
* Chronic or relapse/remitting hemolytic condition or pre-catheterization hematocrit<30 mg/dl
* Unprotected left main coronary disease with >50% stenosis;
* Platelet count <150,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-09

PRIMARY OUTCOMES:
Number of patients who require a vascular groin ultrasound or abdominal CT.
Record occurrence of pseudoaneurysm, arteriovenous fistula, retroperitoneal hematoma, or femoral vein or arterial thrombosis
Record presence of hematoma and size if applicable.
Record hemoglobin drop >3g/dl with over bleeding. Also, record any red cell transfusion due to catheterization related bleeding.

SECONDARY OUTCOMES:
Comparison of time to ambulation.
Occurrence of major and minor bleeding peri-catheterization.
Observe incidence of thrombocytopenia post catheterization defined as a platelet count <100,000.

CONTACTS AND LOCATIONS:
Overall Officials: Herman K Gold, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States